CLINICAL TRIAL: NCT02728687
Title: A Double Blind, Randomized Crossover Study of Efficacy and Safety of Topical Menthol, With and Without Mannitol, in the Treatment of Painful Diabetic Peripheral Neuropathy
Brief Title: Topical Menthol +/- Mannitol for Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Helene Bertrand, MD, CCFP, Clinical instructor, Department of family practice University of British Columbia, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M for PDPN
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: peripheral neuropathy; Diabetes; Pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetes Mellitus; Pain | interventions — Mannitol; Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mannitol and menthol cream (Experimental): Mannitol and menthol cream (Water, Mannitol, Propylene glycol, Isopropyl palmitate. Caprylic capric triglyceride, Ceteareth 20, Cetearyl alcohol, Glyceryl stearate, Polyethylene glycol 100 Stearate, Dimethicone, Octyldodecanol, Menthol, Lecithin, Ethylhexyl glycerin, Phenoxyethanol) applied as needed, up to 4 times daily for one month, to the feet of a person suffering from painful diabetic peripheral neuropathy. During the other month, the menthol cream will be applied to the participant's feet. Whether the mannitol and menthol cream will be given in the first or the second month will be chosen at random. At the end of the 2 months, if the participant chooses this cream, they will be given 3 months' supply of the cream to apply as needed to both feet.
  Interventions: Drug: Mannitol; Drug: Menthol
- Menthol cream (Active Comparator): Cream containing menthol (Water, Propylene glycol, Isopropyl palmitate. Caprylic capric triglyceride, Ceteareth 20, Cetearyl alcohol, Glyceryl stearate, Polyethylene glycol 100 Stearate, Dimethicone, Octyldodecanol, Menthol, Lecithin, Ethylhexyl glycerin, Phenoxyethanol) applied as needed, up to 4 times daily for one month, to the feet of a person suffering from painful diabetic peripheral neuropathy. During the other month, the mannitol and menthol cream will applied to the participant's feet. Whether the menthol cream will be given in the first or the second month will be chosen at random. At the end of the 2 months, if the participant chooses this cream, they will be given 3 months' supply of the cream to apply as needed to both feet.
  Interventions: Drug: Menthol

INTERVENTIONS:
Drug: Mannitol — Apply cream as needed up to 4 times daily to the painful foot and leg
  Other Names: QR cream
  Arms: Mannitol and menthol cream
Drug: Menthol — Apply cream as needed up to 4 times daily to the painful foot and leg

SUMMARY:
Treatments for painful diabetic peripheral neuropathy (PDPN) are not very effective and have multiple side effects. To find out if a menthol cream alone or with added mannitol treats PDPN effectively, 90 participants with PDPN, after one month of observation, will receive randomly assigned menthol cream or the same cream with mannitol added for 3 months with a crossover for 3 additional months. At time 0, 1,4 and 7 months their BPI pain severity and interference scores, DN4 scores, cream % effectiveness and side effects will be compared.

DETAILED DESCRIPTION:
Purpose: to find out if a menthol cream containing mannitol is more effective than the same cream without mannitol in relieving painful diabetic peripheral neuropathy (PDPN). The test cream which will, at a later date, be marketed as QR cream contains Water, Mannitol, Propylene glycol, Isopropyl palmitate. Caprylic capric triglyceride, Ceteareth 20, Cetearyl alcohol, Glyceryl stearate, Polyethylene glycol 100 Stearate, Dimethicone, Octyldodecanol, Menthol, Lecithin, Ethylhexyl glycerin, Phenoxyethanol. The control cream contains the same ingredients minus the mannitol.

Hypothesis: a menthol cream containing mannitol is more effective at relieving the pain, the physical limitations and the emotional distress caused by PDPN than the same cream without mannitol.

Justification: PDPN is common and can be disabling because of the intensity of the pain it can cause. Less than 50% of those suffering from this condition get adequate pain relief from their current medications. The oral medications, anticonvulsants, antidepressants, NSAIDS, marijuana derivatives and narcotics have numerous side effects and are potentially addictive. Topical local anaesthetics have short-lived effect over only a small area and topical capsaicin often causes burning on application and prolonged use destroys the affected nerves. A previous study has demonstrated mannitol's effectiveness in down regulating the capsaicin receptor which is believed to cause the burning sensation of PDPN. A cream containing mannitol has few side effects, and, if effective, may decrease the need for other, more dangerous medications.

Objectives: to show that a menthol cream containing mannitol is more effective, over a period of 28 weeks, than the same cream without mannitol at relieving the pain, the physical limitations and the emotional distress caused by PDPN.

Research Design: this is a randomized, double-blind, placebo-controlled crossover trial involving 3 visits.

Participants who are taking medications or insulin to treat diabetes will have on/off vibration test on the hallux of each foot. If at least 5 of their 8 vibration tests are erroneous or "I don't know", their score on the DN4 questionnaire is >4/10 they will be enrolled.

After 1 month's observation period, 90 participants will be given either a menthol cream with mannitol or the same cream without mannitol to apply to their feet for 3 months, following which the creams will be crossed over for an additional 3 months. Which cream is to be applied in the first 3 months will be chosen at random. Participants and clinicians will be blinded as to cream assignment for the duration of the study. Participants will be instructed to rub the cream on their feet and the tender nerves supplying their feet, 2 to 4 times daily, as needed for pain relief.

At 0,1,4 and 7 month, their BPI pain severity and interference scores, DN4 scores, cream % effectiveness and side effects will be recorded. At 4 and 7 months, they will be compared.

Statistical Analysis: primary endpoint, BPI pain interference scores (how much pain interferes with function and relationships) . t-tests will compare the difference between the maximum daily pain interference score for the menthol cream as compared with the mannitol and menthol cream at 4 and 7 months. Secondary endpoints: BPI pain severity score and DN4 score (how many symptoms of peripheral neuropathy are registered), % cream effectiveness, incidence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* • 19 years of age or older
* Are currently being treated for diabetes with medications or insulin
* Suffering from painful diabetic peripheral neuropathy affecting their feet for at least three months.
* Maximum daily pain or discomfort score in each foot greater than or equal to 5/10.
* Score on the DN4 questionnaire at least 4/10
* At least 5 incorrect or I don't know responses to 8 on/off vibration tests
* Able and willing to attend Dr. Helene Bertrand's office three times.

Exclusion Criteria:

* • Known Allergies to any of the ingredients of the cream
* Open lesions diabetic foot ulcers or abrasions on the skin where the cream will be applied
* Unwilling to stop using other topical products (creams or patches) for the treatment of their neuropathic pain at least 14 days before joining this study.
* Pain in each foot which varies by more than 2/10 from day-to-day
* Pregnant (a urine pregnancy test will be done on women younger than 50 at their first visit )
* breast-feeding,
* Women of reproductive age and not using the following methods of contraception:

  1. Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (DepoProvera, Lunelle), or hormone implant (Norplant System)
  2. Double-barrier method
  3. Non-hormonal intrauterine devices
  4. Vasectomy of partner
* Limited standing or walking from any cause (back, knees, feet, etc) other than diabetic neuropathic pain.
* Giving a history or exhibiting clinical signs of other causes of neuropathic pain such as spinal claudication, severe back pain on standing or walking, or a history of having received chemotherapy.
* Pain extending above the ankles.
* Those with ischemic peripheral vascular disease
* Those receiving acupuncture or using a TENS machine Those undergoing hydrotherapy
* Those who are unable to understand English, French, or Spanish and can not attend Dr. Bertrand's office with someone who will translate for them.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
BPI pain interference improvement 3 months | 3 month
  Compares the change in BPI pain interference score after 3 months of cream use for menthol and mannitol cream and menthol cream alone.

SECONDARY OUTCOMES:
Maximum BPI pain severity improvement 3 months | 3 months
  Compares the change in maximum BPI pain severity score after 3 months of cream use for menthol and mannitol cream and menthol cream alone.
NH4 improvement 3 month | 3 months
  Compares the change in NH4 score after 3 months of cream use for menthol and mannitol cream and menthol cream alone.
% improvement from cream use | 3 months
  Compares the % improvement from cream use after 3 months of cream use for menthol and mannitol cream and menthol cream alone.
Satisfaction score | 3 months
  Compares the Satisfaction score from cream use after 3 months of cream use for menthol and mannitol cream and menthol cream alone.
incidence of side effects | 3 months
  Compares the incidence of side effects from cream use after 3 months of cream use for menthol and mannitol cream and menthol cream alone.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Private Physician's Office, Courtenay, British Columbia
  - Okanagan Interventional Pain Clinic,, Kelowna, British Columbia
  - Suite 303 - 570 Raymer Avenue, Kelowna, BC, Canada, V1Y 4Z5, Nelson, British Columbia
  - Dr. Helene Bertrand Inc., 220-1940 Lonsdale Ave., North Vancouver, British Columbia
  - Maple Tree Medical Clinic, Salmon Arm, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
Age, sex, pain medications used, brief pain inventory pain interference and pain severity scores (BPI), DN4 (neuropathy questionnaire), % effectiveness and side effects of cream.
  An encrypted, de-identified database containing this information will be shared with other researchers when the database is complete.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: As of April 15, 2019, 50 of the 90 participants have been entered into the study. At this rate, the study database should be completed by December 2020.
Access Criteria: University affiliation. Peripheral neuropathy publication.

REFERENCES:
- [Background] Bertrand H, Kyriazis M, Reeves KD, Lyftogt J, Rabago D. Topical Mannitol Reduces Capsaicin-Induced Pain: Results of a Pilot-Level, Double-Blind, Randomized Controlled Trial. PM R. 2015 Nov;7(11):1111-1117. doi: 10.1016/j.pmrj.2015.05.002. Epub 2015 May 12. PMID 25978942
- [Background] Daousi C, MacFarlane IA, Woodward A, Nurmikko TJ, Bundred PE, Benbow SJ. Chronic painful peripheral neuropathy in an urban community: a controlled comparison of people with and without diabetes. Diabet Med. 2004 Sep;21(9):976-82. doi: 10.1111/j.1464-5491.2004.01271.x. PMID 15317601
- [Background] Young MJ, Boulton AJ, MacLeod AF, Williams DR, Sonksen PH. A multicentre study of the prevalence of diabetic peripheral neuropathy in the United Kingdom hospital clinic population. Diabetologia. 1993 Feb;36(2):150-4. doi: 10.1007/BF00400697. PMID 8458529
- [Background] Duby JJ, Campbell RK, Setter SM, White JR, Rasmussen KA. Diabetic neuropathy: an intensive review. Am J Health Syst Pharm. 2004 Jan 15;61(2):160-73; quiz 175-6. doi: 10.1093/ajhp/61.2.160. PMID 14750401
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Perkins BA, Olaleye D, Zinman B, Bril V. Simple screening tests for peripheral neuropathy in the diabetes clinic. Diabetes Care. 2001 Feb;24(2):250-6. doi: 10.2337/diacare.24.2.250. PMID 11213874